CLINICAL TRIAL: NCT00271297
Title: Effect of Pelvic Floor Muscle Training (PFMT) in Prevention and Treatment of Female Pelvic Organ Prolapse (POP).
Brief Title: Pelvic Floor Muscle Training (PFMT) in Treatment and Prevention of POP (POP Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); The Norwegian Women´s Public Health Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-05146; 200501371 SM/RH (NSD)
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Uterine Prolapse; Bladder Diseases; Cystocele; Rectocele
Keywords: pelvic floor; exercise therapy; prevention; ultrasonography; risk factors
MeSH Terms: conditions — Uterine Prolapse; Urinary Bladder Diseases; Cystocele; Rectocele

INTERVENTIONS:
Behavioral: Pelvic floor muscle training

SUMMARY:
Background:

The pelvic floor muscles (PFM) are located inside the pelvis, surrounding the urethra, vagina and rectum. They provide structural support for the pelvic organs. Dysfunctional PFM can lead to urine and fecal incontinence, pelvic organ prolapse (POP), sexual problems and chronic pain syndromes. POP increases with age, parity and weakness in the PFM. Symptoms associated with POP are backache, bladder, bowel and sexual dysfunction, and pelvic heaviness. Thus the condition is debilitating and can greatly affect the quality of life, interfering with day-to-day activities and reduce participation in physical activity.

The aim of the project:

As life expectancy increases, more women may experience POP. Hence it is important to prevent and treat the condition at an early stage. Despite being a common disorder among women, little research has been done on POP. The aim of this study is to evaluate the effect of pelvic floor muscle training (PFMT). PFMT is a non-invasive method with no adverse effects. If there is significant effect, the main goal is to incorporate this method in clinical practice among physiotherapists and medical doctors. If PFM training is effective, more emphasis of PFM training can be put into regular female fitness programs. The prevalence of POP increases with age.

Method:

This is a single blind randomised controlled trial to evaluate the effect of PFMT on POP. 100 women with POP will be randomised to either training or control group. The training programme will last for six months, training once a week with a physiotherapist in addition to a structured home training programme. A blinded case-control study will also be carried out. 50 women without POP will be matched for age and vaginal deliveries. Before starting the RCT study, a reproducibility study on perineal ultrasound will be carried out in 18 women.

DETAILED DESCRIPTION:
Background for the study:

The incidences and prevalence of POP is difficult to determine, since many women do not seek medical advice and treatment for the condition. It has been estimated that half of women who have given birth lose some of the pelvic floor support, resulting in some degree of prolapse. Of these 10-20% will seek medical help. About 10% of all women will at one point in life undergo surgery for a prolapse condition. The incidence of POP requiring surgery after a hysterectomy is 3.6% per 1,000 women per year in the UK.

Treatment of POP can be conservative (PFMT), mechanical (use of a pessary) or surgical. A recently published Cochrane review concluded that there are no studies evaluating the effect of PFMT on POP. PFMT is without adverse effects, and theoretical knowledge of anatomy and function of the PFM provides a basis for trying strength training of the PFM both to prevent and to reverse POP.

In Norway Bø (1990, 1999) PhD, physiotherapist and professor at the Norwegian School of Sport Sciences (NSSS), has developed a training model for strengthening the PFM. The results from several randomised controlled trials of this program have shown high cure and improvement rates both in prevention and treatment of urinary incontinence.

Ultrasound and MR examinations have shown that after vaginal delivery the pelvic floor is situated in a lower position than in nullipara. In addition, the pelvic floor of stress urine incontinent (SUI) women is in a lower position than of continent women. DeLancey et al (2003) showed that women with POP generated 43% less maximum force and had more atrophy of the pelvic floor muscles than women without prolapse. One of the main theories explaining the effectiveness of PFMT on SUI includes factors that may change through strength training: increased cross-sectional area of the muscle (muscle volume), neurogen adaptation, imposed viscoelastic properties ("stiffness") of the connective tissue and altered location of the PFM at a higher level in the pelvic cavity. Morphological changes in relation to PFMT have not been examined in RCTs, but have shown a cure rate of 44-70% measured as < 2 gram leakage in various pad tests and significant increase in muscle strength after PFMT.

Several studies have shown that > 30% of women are unable to contract the PFM properly at the first consultation. Bump et al (1991) showed that 25% were pushing downwards instead of lifting up and in. Other common mistakes are to use muscle groups outside the pelvic area instead of the PFM. Instruction, feedback, close follow-up and high adherence are important factors if the strength training.

Objective:

The aim of the present study is to evaluate whether PFMT can reverse and prevent further development of POP. The project comprises a RCT (main study). In addition we will conduct a case-control study to investigate risk factors, such as muscle strength and joint flexibility in women with and without POP. The project description below will focus on the RCT. The same measurements will be used in the case-control study, and women participating in the RCT will be cases of the case-control study.

Method, design:

The main study is a prospective randomised trial. Women with POP will be referred by selected community gynaecologists working in Oslo and Akershus. Those who express an interest in participating in the project will be referred to physiotherapist and manual therapist Ingeborg Hoff Brækken, who is the project manager. The women will participate in a structured interview; complete a questionnaire about symptoms and quality of life and undergo a clinical examination at. Gynaecologist Majida at Akershus university hospital will conduct the ultrasound examination. The women will be stratified by the stage of prolapse after the pelvic floor prolapse quantifying (POPQ). They will then be randomised into two groups; PFMT or control. Brækken will train the intervention group at Hans & Olaf Fysioterapi A/S. The gynaecologist will be blinded for group allocation. After 6 months all women from both groups will be referred to the physiotherapist where they will complete the same questionnaire about symptoms and quality of life and measure PFM strength. The gynaecologist will then conduct the same ultrasound examination and POPQ.

Drop-out routines:

The "intention to treat" principle will be followed. Moreover, a per-protocol analysis will be carried out in those who have completed ≥ 80% of the recommended training regimen.

Protocol for PFMT:

1. Pre-contraction (the "knack"). All women will be taught how to contract the PFM before, during and after increases in abdominal pressure (coughing, sneezing, heavy lifting)
2. Home training. The intervention group will be asked to perform 3 sets of 8-12 near maximum contractions per day in different positions with the legs abducted. All women will receive a booklet and a DVD showing the exercise program. Adherence will be noted in a diary
3. Training and follow-up with a physiotherapist. The women visit the physiotherapist for training with vaginal pressure biofeedback once a week for 3 months. For the next 3 months they train once every second week with the physiotherapist (total of 18 times). Muscle strength is registered at each visit.

The control group receives no treatment. After the project period they will be referred to a physiotherapist if they so wish.

Case-control study:

In parallel with the training intervention, 50 female controls without POP will be referred from the same gynaecologists. In this case-control study only women with stage 0 on POPQ will be included in the control group. They will be examined in the same way as the main study group by the physiotherapist and gynaecologist. PFM strength and clinical tests for "benign hypermobility joint syndrome" will be conducted. They also complete the same forms as in the RCT.

Statistical analysis:

We use SPSS version 11 for data analysis with relevant statistical methods to compare the groups. Results of continuous variables will be given as an average of 95% CI. Results will be given as numbers needed to treat (NNT). The level of significance will be set at < 5%. Professor of statistics, Ingar Holme PhD, NSSS, is advising the project.

Ethics

Names and personal identity numbers will not be registered. All data will be stored in a locked and fireproof cabinet. Data is filed in the same way as all the project data at Norwegian Social Sciences Data Services (NSD) in Bergen. The project complies with the Helsinki declaration in requiring all participants to give their written informed consent. The project has been approved by the Southern Regional Health Authority's committee on medical ethics.

ELIGIBILITY:
Pelvic organ prolapse (POP) is defined as grade 1 or more on POP-Q. This means that the most distal portion of the prolapse is less than 1 cm above the level of the hymen or that the distal edge of the cervix or vaginal cuff (post hysterectomy) is more than 2 cm lower than the total vaginal length.

Inclusion Criteria:

* Parous women in Oslo and Akershus
* POP grade 1-3 on POP-Q.
* Age 18-70

Exclusion Criteria:

* Women with POP-Q grade 0 or 4 and women with cervix elongation
* Women with other disease: radiating back pain, neurological disorders, previous pelvic cancer, psychiatric or other disorders that have an impact on ability to train or the condition (l.o. asthma). Women who is under treatment for cancer or uses muscle relaxants
* Previous POP surgery
* Women who wants to use pessary/ ring during the intervention period and three weeks prior to this
* Pregnant or nursing women, or women planning to become pregnant in the intervention period
* Women with untreated urinary tract infection
* Women who do not understand Norwegian
* Woman planning to be away more than 4 weeks of the intervention period
* Women who cannot contract the PFM

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
RCT:
Localisation of bladder neck, cervix and rectal ampulla at rest (translabial ultrasound)
Subjective symptoms score (Mouritsen and Larsen 2003, Tegerstedt et al in press, Avery et al 2004)
Ultrasound measurement of changes in muscle morphology: 1. thickness of levator ani
Size of levator hiatus
Levator activity during contraction, coughing and Valsava manoeuvre.
Case control study:
Comparison of background variables and risk factors
Presence of "Benign Hypermobility Joint Syndrome"
Measurement PFM strength
Reproducibility study:
Reproducibility of ultrasound examination of localisation and function of PFM and POP (same measurements as in the RCT)

SECONDARY OUTCOMES:
RCT study:
Independent variables (muscle function and strength)is vaginal palpation, visual observation of perineum, measurement of muscle strength with Camtech fibreoptic microtransducer connected to a vaginal balloon(Camtech AS, Sandvika, Norway)
* Training diary for registration of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, Prof, Dr.sci, Study Director — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, department of Sports Medicine, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Hoff Braekken I, Majida M, Engh ME, Bo K. Morphological changes after pelvic floor muscle training measured by 3-dimensional ultrasonography: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):317-324. doi: 10.1097/AOG.0b013e3181cbd35f. PMID 20093905